CLINICAL TRIAL: NCT06176924
Title: Effect of tDCS Along With Relaxation Technique on Anxiety Level in Students Preparing for Competitive Exams: A Randomized Controlled Trail
Brief Title: Effect of tDCS Along With Relaxation Technique on Anxiety Level in Students Preparing for Competitive Exams
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Subhasish Chatterjee, Effect of tDCS along with relaxation technique on anxiety level in students preparing for competitive exams: A Randomized Controlled Trial, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPC-PA-06
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Anxiety
Keywords: Anxiety, tDCS, Relaxation, Competitive Exam Students, 2mA, CSAI-2R
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation; Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS and Relaxation technique (Experimental): Subjects within an experimental group had received 9 sessions of tDCS (2mA, 20 min anode placed on DLFPC of left side and cathode on supraorbital cortex of right side) along with relaxation technique.
  Interventions: Device: tDCS; Other: Relaxation technique
- Relaxation technique (Other): Subjects in the control group are going to receive 9 sessions of relaxation technique
  Interventions: Other: Relaxation technique

INTERVENTIONS:
Device: tDCS — tDCS (2mA, 20 min anode placed on DLFPC of left side and cathode on supraorbital cortex of right side) along with relaxation technique.
  Arms: Active tDCS and Relaxation technique
Other: Relaxation technique — Relaxation technique

SUMMARY:
Anxiety is one of the most significant obstacles to academic success. When stress is interpreted negatively or becomes overwhelming, it causes anxiety before and during examinations, which in turn impacts students' academic performance. The difficulty in managing severely associated anxiousness enhances the demand for NIBS. It is a unique approach that has the potential to alleviate anxiety by modifying cortical excitability whereas Relaxation breaks the vicious cycle of pain caused by muscular stress, circulatory illness, and metabolic by-products alterations. The main purpose is to evaluate whether tDCS along with Relaxation technique reduces the anxiety level in competitive exam students. Total 46 students are recruited and randomly allocating in experimental and control group. The subjects in the experimental group are going to receive 9 tDCS sessions (2mA, anode placed on the DLFPC of left side and cathode on right supraorbital cortex for 20 min) along with relaxation technique. Subjects in the control group are going to receive 9 sessions of relaxation. The CSAI-2R scale is used as an Outcome Measure. Samples completed the CSAI-2R scale before and following the intervention. The data will be analyzed using SPSS 26.0 software.

ELIGIBILITY:
Inclusion Criteria: • Both male and female students.

* Competitive Exam students only.
* Age group between 15 years to 18 years.
* Willingness to take part in the research.

Exclusion Criteria: • Seizure disorder

* Non-Corporative students
* Skin irritation

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
CSAI- 2R (Competitive State Anxiety Inventory-2R) | 5 minutes
  It is a reliable and viable scale for assessing the level of competitive anxiety. It's having 27 components, each having 4 grades ranging from 1 to 4.

CONTACTS AND LOCATIONS:
Locations (1):
- MMIPR, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No